CLINICAL TRIAL: NCT00123773
Title: A Phase II Study of F-Fluorodeoxyglucose (FluGlucoScan) in Patients With Known or Suspected Cancers of Low Incidence
Brief Title: Study of F-Fluorodeoxyglucose (FluGlucoScan) in Patients With Known or Suspected Cancers of Low Incidence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SP-14-0038/DX-FDG-003/21386; NCT00271648 (obsolete NCT alias)
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-03

CONDITIONS: Sarcoma; Multiple Myeloma; Testicular Neoplasms; Ovarian Neoplasms; Kidney Neoplasms
Keywords: positron emission tomography; fluorodeoxyglucose F18; Tomography scanners, x-ray computed
MeSH Terms: conditions — Sarcoma; Multiple Myeloma; Testicular Neoplasms; Ovarian Neoplasms; Kidney Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Positron Emission Tomography

SUMMARY:
Positron Emission Tomography (PET) is a specialised nuclear medicine procedure that uses positron emitting radiolabeled tracer molecules to measure biological activity. The most common of these radiolabeled tracers is 18F-fluorodeoxyglucose (18F-FDG), which is used to determine abnormal glucose metabolism in tumours and other sites. It has general applications in all areas where abnormal glucose metabolism may be present including in circumstances such as differentiating the tumour from scar tissue; evaluating the presence of the tumour in light of rising tumour markers and normal morphological imaging techniques; and assessing response to therapy where other techniques are deemed to be unhelpful. The Cross Cancer Institute has recently been funded to establish a PET centre, and this study will evaluate the effectiveness, value and safety of PET scanning in a number of uncommon cancers in the Canadian health care environment.

DETAILED DESCRIPTION:
Background

Positron Emission Tomography (PET) is a specialised nuclear medicine procedure that uses positron emitting radiolabeled tracer molecules to measure biological activity. The most common of these radiolabeled tracers is 18F-fluorodeoxyglucose (18F-FDG), which is used to determine abnormal glucose metabolism in tumours and other sites. It has general applications in all areas where abnormal glucose metabolism may be present including in circumstances such as differentiating the tumour from scar tissue; evaluating the presence of the tumour in light of rising tumour markers and normal morphological imaging techniques; and assessing response to therapy where other techniques are deemed to be unhelpful.

The Cross Cancer Institute has recently been funded to establish a PET centre that will establish a research programme to prove the effectiveness of PET scanning in the Canadian health care environment and validate the data that have been developed in other jurisdictions in specific oncologic indications.

Objectives

Primary Objective - The objective of the clinical trial is to establish the general utility and value of 18F-FDG PET imaging in patients with known or suspected myeloma, sarcoma, testicular cancer (seminomatous and non-seminomatous germ cell tumors), endometrial cancer, ovarian cancer, cervical cancer, transitional cell carcinoma of the bladder, renal cell carcinoma, pancreatic, adenocarcinoma, mesothelioma and gastric cancer.

Secondary Objectives - The secondary objective of the clinical trial is to demonstrate the safety by documentation of adverse events.

Study Design

The proposed clinical trial will be a Phase II, diagnostic imaging, open label, single site, clinical trial in patients with defined oncologic disease. The patient population will consist of patients with suspected or known infrequently occurring cancers, which are not covered by Protocol DX-FDG-001. This population includes patients with known or suspected myeloma, sarcoma, testicular cancer (seminomatous and non-seminomatous germ cell tumors), endometrial cancer, ovarian cancer, cervical cancer, transitional cell carcinoma of the bladder, renal cell carcinoma, pancreatic adenocarcinoma, mesothelioma and gastric cancer.

Each patient will receive a single IV injection of 18F-FDG. Imaging will be conducted 60 minutes after an average injection of 200 - 300 MBq of 18F-FDG in hydrated, fasted patients. Images will be collected for 40 to 60 minutes in 5 - 7 body positions (total counts 5 to 15 million) using either the C-PET, Allegro or Gemini PET scanners located in Nuclear Medicine. Standard transaxial images will be reconstructed from the collected data and can be re-oriented into coronal or sagittal slices as required. The images will then be examined by an experienced nuclear medicine physician with regard to normal physiological uptake of 18F-FDG. The location and intensity of abnormal 18F-FDG uptake will be noted and correlated with clinical findings, and conventional imaging techniques, as available.

Statistical Analyses

Sample Size

The study will enrol approximately 220 subjects, with an approximate maximum of 20 subjects per specific tumour type (myeloma, sarcoma, testicular cancer [seminomatous and non-seminomatous germ cell tumors], endometrial cancer, ovarian cancer, cervical cancer, transitional cell carcinoma of the bladder, renal cell carcinoma, pancreatic adenocarcinoma, mesothelioma and gastric cancer).

Statistical Analyses

For each group, the investigators will calculate the positive predictive value (true positive outcomes/true positive outcomes + false positive outcomes) of the 18F-FDG scan. They also intend to evaluate the percentage of patients in which the 18F-FDG outcome affected patient management.

Criteria for Evaluability of Study Subject Data

All subjects receiving 18F -FDG will be evaluated for safety and efficacy.

Study Population

Number of Subjects to be Studied

Approximately 220 patients overall; approximately 20 in each cancer type.

Inclusion Criteria for Selection of Study Subjects

Patients will be included in the study if they meet all of the following criteria.

1. Male or female. If female of child-bearing potential and outside of the window of 10 days since the last menstrual period, a negative serum pregnancy test.
2. Known or suspected primary or metastatic tumours of myeloma, sarcoma, testicular cancer (seminomatous and non-seminomatous germ cell tumors), endometrial cancer, ovarian cancer, cervical cancer, transitional cell carcinoma of the bladder, renal cell carcinoma, pancreatic adenocarcinoma, mesothelioma and gastric cancer.
3. Age greater than or equal to 15 years.
4. Able and willing to follow instructions and comply with the protocol.
5. Provide written informed consent prior to participation in this study.

7. Karnofsky Performance Scale score 60 - 100.

Exclusion Criteria

Patients will be excluded from the study if they meet any of the following criteria:

1. Having had surgery or radiotherapy within 10 days of the planned imaging study.
2. Nursing or pregnant females.
3. Age less than 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. (If female of child bearing potential and outside of the window of 10 days since the last menstrual period, a negative serum or urine pregnancy test is required.)
* Known or suspected primary or metastatic tumours of myeloma, sarcoma, testicular carcinoma (seminomatous and non-seminomatous germ cell tumours), endometrial carcinoma, renal cell carcinoma, pancreatic adenocarcinoma, malignant mesothelioma, gastric carcinoma and cholangiocarcinoma.
* Age equal to or greater than 15 years
* Able and willing to follow instructions and comply with the protocol
* Provide written informed consent prior to participation in this study
* Karnofsky Performance Scale score 60-100

Exclusion Criteria:

* Nursing or pregnant females
* Having had surgery or radiotherapy within 10 days of the planned imaging study
* Presence of a severe infection
* Age less than 15 years
* Blood glucose greater than 10mmol/L

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2004-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To confirm the diagnostic effectiveness of 18F-FDG in patients with known or suspected carcinoma

SECONDARY OUTCOMES:
To determine the clinical relevance of PET scans within these patient groups

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McEwan, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada